CLINICAL TRIAL: NCT03445611
Title: Clinical Significance of Parabens Flocculation on the Anti Inflrammmatory Effects of Corticosteroid Injection Osteoarthritic Knees
Brief Title: Parabens Flocculation on the Anti Inflammatory Effects of Corticosteroid Injections for Total Knee Arthroplasty
Acronym: 5160373
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: IRB process never completed.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5160373
Record Dates: First submitted 2017-10-19; First posted 2018-02-26 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Masking Description: randomized into either Group1 or Group 2 medication with or without presevatives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): These patients will receive a corticosteroid solution with lidocaine containing parabens.
  Interventions: Drug: corticosteroid solution with lidocaine containing parabens.
- Group 2 (Active Comparator): These patients will receive corticosteroid solution with paraben free lidocaine.
  Interventions: Drug: corticosteroid solution with lidocaine containing no paraben

INTERVENTIONS:
Drug: corticosteroid solution with lidocaine containing parabens. — To identify whether corticosteroid use with anesthetics containing parabens reduces clinical effectiveness relative to para-free preparations.
  Arms: Group 1
Drug: corticosteroid solution with lidocaine containing no paraben — To identify whether corticosteroid use with anesthetics containing parabens reduces clinical effectiveness relative to para-free preparations.
  Arms: Group 2

SUMMARY:
The purpose of this study is to identify whether corticosteroid use with anesthetics containing preservatives (parabens) reduces clinical effectiveness of the anti-inflammatory agent Up to 100 patients, both male and female, between the ages of 18-89 will be enrolled and randomized into either of the following groups; Group 1: These patients will receive a corticosteroid solution with lidocaine containing parabens.

Group 2: These patients will receive corticosteroid solution with paraben free lidocaine.

DETAILED DESCRIPTION:
Corticosteroid injections have been used to treat inflammatory conditions for many decades (Storz 1973; Roszental, Zurakowski and Blazar 2008). In order to maximize the effectiveness on the synovial tissue, the concentrated form of corticosteroids is typically mixed with an anesthetic preparation. The corticosteroid suspension in a large volume of anesthetic can then disperse throughout the entire joint more effectively, especially in larger joints such as the knee (Centeno and Moore 1994). In addition, the anesthetic provides immediate relief to the area and can help verify that the injected site was the source of pain (Cole and Schumacher 2005). Typical preparations of anesthetic medications are sold in multi-use vials. The anesthetic solution usually contains a paraben preservative, except in the single vials used for spinal injections, because the use of paraben preservatives is contraindicated in spinal injections (Centeno and Moore 1994).

Celestone and Kenalog are two corticosteroid products that are commonly used for intra-articular injections. If co-administration of a local anesthetic is desired, the suspension of Celestone or Kenalog is commonly mixed with 1% or 2% Lidocaine hydrochloride from multi-use vials containing parabens in Orthopedic and Rheumatology clinics.

The orthopedic literature relating to injections rarely addresses the use of the anesthetic commonly used in injections. Flocculation occurs significantly when parabens are present, but the influence on the efficacy of the corticosteroid is unknown (Philipose et al. 2011; Hwang et al. 2016). There is abundant evidence that flocculation occurs when steroids are mixed with anesthetic solutions containing parabens however, the clinical significance of this phenomenon has not been reported. (Skedros and Pitts 2008b; Andreson, Deodhar and O'Rourke 2005; Skedros and Pitts 2008; Lutt, O'Rouke and Deodhar 2007; Cole and Schumacher 2005).

Cole and Schumacher (2005) suggest that flocculation can result from a chemical incompatibility between corticosteroid and other agents. Flocculation that occurs when corticosteroid is mixed with an anesthetic containing parabens may reduce the anti-inflammatory effect of the steroid. There are two possible mechanisms in which the corticosteroid preparation may be less effective. Flocculation may cause the corticosteroid to precipitate, thus reducing dispersal within the injected area (Centeno and Moore 1994). Additionally, flocculation may result from corticosteroid bonding with another molecule (such as methylparaben) within the anesthetic preparation, making it chemically less effective. The purpose of this study is to identify whether corticosteroid use with anesthetics containing parabens reduces clinical effectiveness relative to paraben-free preparations.

STUDY DESIGN:

OBJECTIVES:

The purpose of this study is to identify whether corticosteroid use with anesthetics containing parabens reduces clinical effectiveness relative to para-free preparations.

Hypothesis Alternate: Flocculation due to lidocaine containing parabens decreases the anti-inflammatory effects of corticosteroids when compared to paraben-free lidocaine.

Procedure:

The investigator will enroll up to 100 patients, both male and female, between the ages of 18-89. Once the patient has been consented, They will be randomized into group 1 or group 2. The randomization is a 1 to 1 ratio. Subsequent follow-up via phone call will take place on week 1, week 2, week 4, week 8, and week 16.

Group 1: These patients will receive a corticosteroid solution with lidocaine containing parabens.

Group 2: These patients will receive corticosteroid solution with paraben free lidocaine.

Corticosteroid injections will be given with or without ore-aspiration of synovial fluid. Patient will be in supine position with superior-lateral injection.

Material identification: Celestone soluspan or Kenalog 1% 50mL multiuse vials without epinephrine, 1% 5mL lidocaine vials, 10mL syringes with 21mm x 1 ¼ inch needles, alcohol swabs, exam gloves, betadine solution.

DATA COLLECTION:

The investigator will collect the patients age, sex, BMI, Medical history, along with the WOMAC survey, which asks about the patients knee and activity level and VAS, pain sale (0-10) 0 being the lease amount of pain and 10 being the worst.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of symptomatic primary knee osteoarthritis according to the American Rheumatism Association classification criteria for knee osteoarthritis, ability to understand study protocol and agreement to participate

Exclusion Criteria:

* History of any knee injection in the past 6 months, History of more than 2 injections in the knee under study, previous fracture or surgical procedure of knee under investigation, any benign or malignant tumor in knee, chemotherapy, hemearthosis, current infection in the affected limb.

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2019-10-15 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
WOMAC-Western Ontario and McMaster Universities Osteoarthritis Index | 6 months
  This is a survey that asks your view about your knee. This information will help track how you feel about your knee and how well you are able to do your usual activities

SECONDARY OUTCOMES:
VAS-Visual Analogue Scale | 6 months
  This is a Scale used to measure pain intensity. It is a continuous scale comprised of a horizontal line, usually 10cm or 100mm in length, the patient will mark a line between the two end-points, indicating there pain level.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Health, Department of Orthopaedic Surgery, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Undecided